CLINICAL TRIAL: NCT01328964
Title: Comparison of Asthma-related Outcomes and Costs in Pediatric Subjects That Received Fluticasone Propionate, Budesonide or Montelukast in a Large Managed Care Population
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112608
Record Dates: First submitted 2010-03-04; First posted 2011-04-05 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: pediatric; asthma; outcomes; inhaled cortcosteroids
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Budesonide; Commerce; montelukast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children Ages 4-11 with asthma: Children ages 4 to 11 with a diagnosis of asthma receiving a prescription for an asthma therapy
  Interventions: Drug: Fluticasone propionate; Drug: Budesonide; Drug: Montelukast

INTERVENTIONS:
Drug: Fluticasone propionate — fluticasone propionate 44 mcg
  Other Names: Flovent® is a registered trademark of GlaxoSmithKline
Drug: Budesonide — budesonide
  Other Names: Singulair®is a registered trademark of Merck and Company
Drug: Montelukast — montelukast
  Other Names: Rhinocort® is a registered trademark of AstraZeneca

SUMMARY:
The objective of this study is to compare asthma-related exacerbations (emergency department (ED) or inpatient (IP) visit) and related cost in pediatric patients aged 4-11 years that received either fluticasone propionate 44 mcg (FP44) or budesonide (BUD) or montelukast (MON). This retrospective observational cohort analysis utilizes a large managed care database with linked pharmacy and medical claims. Patients with ≥ 1 pharmacy claim FP44 or BUD or MON between January 1, 2000 through June 30, 2008 (4-11 years old at time of index) with ≥ 1 diagnosis for asthma (ICD-9 493.xx) in the pre-index period and continuously eligible to receive healthcare services for 1-year pre-index and at least 30 days post-index. Dose of each inhaled corticosteroid was not known in the database. Follow-up was defined for each patient as the period beginning with the index date and ending with the last date of continuous claims history, switch to another asthma controller medication, or claim for an asthma related event (ED/IP visit or OCS use) post-index, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* ICD-9 code for asthma
* one or more outpatient pharmacy claims for fluticasone propionate 44mg or budesonide between January 1, 2000 and June 30, 2008
* ages 4 to 11 years

Exclusion Criteria:

* diagnosis of Cystic Fibrosis
* ≥ 1 Rx claim for any asthma controller in the pre-index period

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Claims related to pediatric patients age 4-12 in the database with one or more outpatient pharmacy claims for fluticasone propionate 44 micrograms (FP44) or budesonide (BUD) or montelukast (MON) between January 1, 2000 and June 30, 2008.
Sampling Method: Non-Probability Sample
Enrollment: 9906 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective observational study utilizing a large managed care database with linked pharmacy and medical claims. The dose of each inhaled corticosteroid was not known in the database.
Groups:
- Fluticasone Propionate: Pediatric participants aged 4-11 years that received fluticasone propionate 44 micrograms (FP44) for the treatment of asthma
- Budesonide: Pediatric participants aged 4-11 years that received budesonide for the treatment of asthma
- Montelukast: Pediatric participants aged 4-11 years that received montelukast for the treatment of asthma
Period: Overall Study
Arm/Group | Fluticasone Propionate | Budesonide | Montelukast
Started | 2212 | 3270 | 4424
Completed | 2212 | 3270 | 4424
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate | Budesonide | Montelukast | Total
Number analyzed (Participants) | 2212 | 3270 | 4424 | 9906
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.18 (2.20) | 7.30 (2.27) | 7.21 (2.23) | 7.23 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 897 | 1267 | 1797 | 3961
  Male | 1315 | 2003 | 2627 | 5945

OUTCOME MEASURES:

1. Primary Outcome: Number of Asthma-related Hospitalizations, Asthma-related Emergency Department (ED) Visits, and Combined Hospitalizations/ED Visits Represented Per 100 Person Years
Description: The number of participants with an asthma-related event was computed during the follow-up period and was standardized by dividing by the total days of follow-up in each cohort since participants had different lengths of follow-up. Per 100 person years is equal to the percent of events that occurred during the observed time period of the study.
Time Frame: January 1, 2000 to June 30, 2008
Population: Members of the IMS Life Link Health Plans Claims Database (containing data from >=90 managed healthcare plans, encompassing >=60 million lives) who had >=1 pharmacy claim during the study period. FSC participants were matched 1:2 to budesonide and montelukast separately, leading to different numbers analyzed for FSC dependent on cohort of interest.
Measure: Number; unit: asthma events per 100 person years
Arm/Group | Fluticasone Propionate | Budesonide
Number analyzed (Participants) | 1635 | 3270
asthma events per 100 person years
  Hospitalizations | 0.89 | 0.61
  Emergency Department Visits | 3.35 | 5.30
  Hospitalizations or Emergency Department Visits | 4.17 | 5.85
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Budesonide; Test type: Superiority or Other; p < 0.0001, Regression, Cox — The p-value is a comparison of the combined hospitalization/emergency department visit endpoint; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.51 to 0.974]

2. Secondary Outcome: Mean Monthly Asthma-related Costs (Pharmacy and Medical) During the Post-index Period
Description: The mean total asthma costs are a sum of pharmacy and medical costs. Costs were determined monthly from the pharmacy and medical encounters recorded in the managed care insurance database. All costs were summed for each participant over the 3-12 month follow-up period (post-index period), and a mean monthly cost was calculated by dividing by the follow-up for each participant.
Time Frame: 12 months prior to January 1, 2000 to June 30, 2008
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Fluticasone Propionate | Budesonide
Number analyzed (Participants) | 1635 | 3270
United States dollars
  Monthly Medical Costs | 25 (126) | 27 (166)
  Monthly Pharmacy Costs | 20 (40) | 32 (71)
  Monthly Total Costs | 45 (136) | 59 (186)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Budesonide; Test type: Superiority or Other; p < 0.001, Regression, Linear — P-value is based on the differences in the total monthly asthma costs; Mean Difference (Net) = -14, 95% CI 2-sided [-19 to -9]

3. Secondary Outcome: Number of Asthma-related Hospitalizations, Asthma-related Emergency Department (ED) Visits, and Combined Hospitalizations/ED Visits Represented Per 100 Person Years
Description: as for outcome 1
Time Frame: 12 months prior to January 1, 2000 to June 30, 2008
Population: as for outcome 1
Measure: Number; unit: Asthma related events per100 person year
Arm/Group | Fluticasone Propionate | Montelukast
Number analyzed (Participants) | 2212 | 4424
Asthma related events per100 person year
  Hospitalizations | 0.71 | 0.62
  Emergency Department Visits | 3.40 | 4.76
  Hospitalizations or Emergency Department Visits | 4.07 | 5.29
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Montelukast; Test type: Superiority or Other; p = 0.0495, Regression, Cox — P-value is based on the comparison of combined endpoint of hospitalization/emergency department visits; Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.565 to 0.999]

4. Secondary Outcome: Mean Monthly Asthma-related Costs (Pharmacy and Medical) During the Post-index Period
Description: as for outcome 2
Time Frame: 12 months prior to January 1, 2000 to June 30, 2008
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Fluticasone Propionate | Montelukast
Number analyzed (Participants) | 2212 | 4424
United States dollars
  Monthly Medical Costs | 26 (165) | 27 (176)
  Monthly Pharmacy Costs | 21 (87) | 48 (75)
  Monthly Total Costs | 48 (190) | 75 (197)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Montelukast; Test type: Superiority or Other; p < 0.0001, Regression, Linear — P-value is based on difference in total monthly asthma costs; Mean Difference (Net) = -28, 95% CI 2-sided [-28 to -27]

ADVERSE EVENTS:
Description: This was a retrospective observational study utilizing a large managed care database with linked pharmacy and medical claims. Serious adverse events and non-serious adverse events were not collected.
Arm/Group | Fluticasone Propionate | Budesonide | Montelukast
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.